CLINICAL TRIAL: NCT06055023
Title: Phase I Clinical Study on the Tolerability, Safety and Pharmacokinetics of Single-dose Dose Escalation and Multiple-dose Oral ZL-82 Tablets in Healthy Adult Subjects
Brief Title: Phase I Clinical Study of ZL-82 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: H-ZL82-PI-I
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis (RA); Inflammatory Bowel Disease - IBD1
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZL-82 (Experimental): 1 case，The starting dose，Take the medicine once on D1 ，D1 through 7.
  Interventions: Drug: ZL-82 12.5mg; Drug: ZL-82 25mg; Drug: ZL-82 50mg; Drug: ZL-82 100mg; Drug: ZL-82 200mg; Drug: ZL-82 300mg; Drug: ZL-82 450mg; Drug: ZL-82 600mg
- zL-82 placebo group (Placebo Comparator): 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Interventions: Drug: zL-82 placebo 12.5mg; Drug: ZL-82 placebo 25mg; Drug: ZL-82 placebo 50mg; Drug: ZL-82 placebo 100mg; Drug: ZL-82 placebo 200mg; Drug: ZL-82 placebo 300mg; Drug: ZL-82 placebo 450mg; Drug: ZL-82 placebo 600mg

INTERVENTIONS:
Drug: ZL-82 12.5mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 25mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 50mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 100mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 200mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 300mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 450mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: ZL-82 600mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: ZL-82
Drug: zL-82 placebo 12.5mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 25mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 50mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 100mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 200mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 300mg — 1 case,The starting dose,Take the medicine once on D1,D1-7. Edit
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 450mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group
Drug: ZL-82 placebo 600mg — 1 case,The starting dose,Take the medicine once on D1,D1-7.
  Arms: zL-82 placebo group

SUMMARY:
ZL-82 is an oral janus kinase (JAK) inhibitor. In vitro biological mass spectrometry identification test proves that ZL-82 can selectively and irreversibly inhibit JAK3. It has obvious safety advantages, with a wide therapeutic window and controllable cardiotoxicity. This is also demonstrated from preliminary GLP-conditions of acute toxicity in SD rats and Beagle dogs. Results of 4-week long-term toxicity in Beagle dogs also support this notion. Therefore, ZL-82 has the potential to treat rheumatoid arthritis. It Used to relieve and heal swelling, pain, stiffness, and limited mobility that may be caused by rheumatoid arthritis.The drug is intended to be used in patients with RA to relieve and heal swelling, pain, stiffness, and limited mobility that may be caused by rheumatoid arthritis.

Pharmacodynamic studies show that ZL-82 has a strong inhibitory effect on JAK3 with IC50 of 2.8 nM, and has no obvious inhibitory effect on JAK1, JAK2 and TYK2. Compared with the similar drug Tofacitinib, its inhibitory effect on JAK3 subtype is 1nM, but its inhibition IC50 for JAK1 subtype and JAK2 subtype are 112nM and 20nM, respectively.and its selectivity is 100-fold and 20-fold, respectively.Also, the selectivity multiples of ZL-82 were 100-fold and 20-fold than tofacitinib , respectively, which indicates that ZL-82 is more selective than the marketed Tofacitinib.This allows ZL-82 to precisely inhibit JAK kinase and block a series of cytokines in the downstream signaling pathway. And show significant effect on rheumatoid arthritis.

The experimental results showed that in DTH and CIA models, 25, 50, 75, and 100 mg/kg of this variety could dose-dependently inhibit joint swelling in mice.

Objectives of Study

Main Purpose:

1. To evaluate the tolerability, safety and pharmacokinetic characteristics of a single oral dose of ZL-82 tablets in healthy adult subjects;
2. To explore the effect of eating on the PK of oral ZL-82 tablets in healthy adult subjects;
3. To evaluate the tolerability, safety and pharmacokinetics of ZL-82 tablets after multiple oral administration in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, regardless of gender, 18 to 45 years old (including 18 and 45 years old)
* The weighing of male subjects ≥ 50kg, female subjects ≥ 45kg, and a body mass index (BMI) between 19 and 25kg/m2 (including boundary values)
* The medical history, physical examination, laboratory examination items and various tests and tests related to the trial before enrollment were normal or abnormal without clinical significance, and the clinical research doctor judged that they were qualified.
* Be able to understand the informed consent form, voluntarily participate in the trial and sign the informed consent form

Exclusion Criteria:

* Allergic constitution, such as those who are known to be allergic to two or more substances, or those who are known to be allergic to JAK inhibitors or to the excipients contained in the test drug
* ALT and/or AST>1×ULN, TIB>1×ULN, GGT>1×ULN; Scr>1×ULN
* Major surgery within the 3 months prior to the trial or planning to undergo surgery during the trial
* Acute illness within 2 weeks prior to trial
* Have any serious diseases such as cardiovascular system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, malignant tumor, mental illness, etc.
* History of dysphagia or any gastrointestinal disease (or gastrointestinal resection, etc.) affecting drug absorption
* HIV antibody, Treponema pallidum antibody, hepatitis B surface antigen and hepatitis C antibody test are positive
* Positive urine drug screen (including morphine, methamphetamine, ketamine, MDMA, THC)
* Systolic blood pressure>140mmHg or diastolic blood pressure>90mmHg during the screening period;
* Blood donation or blood loss ≥400mL within 3 months, or blood transfusion; blood donation or blood loss ≥200mL within 1 month;
* Have special requirements for diet or cannot comply with the unified diet and corresponding regulations of the research center
* Alcoholics (alcoholism refers to drinking 60-degree white wine ≥10.5L or red wine ≥3.5L per week for more than 5 years), drinking a lot of coffee-containing beverages (more than 8 cups per day, 1 cup = 250ml) or heavy smoking (average > 20 sticks/day);
* Have used any prescription drugs (JAK inhibitors, etc.) that may have an effect on the test drug within 2 weeks;
* 4 weeks (28 days) before enrollment, strong inducers of liver metabolic enzymes was limit. ( such as omeprazole, barbiturates, carbamazepine, aminoglutamine, griseofulvin, carbamazepine, Phenytoin, Gluter, Rifampicin, Sulfinpyrazone, Roxithromycin, etc. )
* Participate in clinical trials of other drugs or medical devices as subjects within 3 months
* Women who are pregnant or breastfeeding or women of childbearing age who have had unprotected sex with their partner within 14 days before the test;
* The subjects or their partners are unwilling to use non-drug contraceptive measures (such as total abstinence, condoms, IUDs, ligation, etc.) for contraception during the trial, or the subject and his partner has a pregnancy plan within 6 months of signing the informed consent;
* Not suitable to participate in the trial according to the judgment of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2023-04-09 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ZL-82：Cmax | 24hours
  Estimation of maximum observed plasma concentration
Pharmacokinetics (PK) of ZL-82：Tmax | 24hours
  Estimation of time to reach Cmax
Pharmacokinetics (PK) of ZL-82：AUC0-24h | 24hours
  Estimation of AUC from time zero to the last measured time point
Pharmacokinetics (PK) of ZL-82：AUC0-∞ | 24hours
  Estimation of AUC from time zero extrapolated to infinity
Pharmacokinetics (PK) of ZL-82：Vd | 24hours
  Estimation of apparent volume of distribution
Pharmacokinetics (PK) of ZL-82：t1/2 | 24hours
  Estimation of terminal elimination half-life
Pharmacokinetics (PK) of ZL-82：CLz/F | 24hours
  Estimation of clearance when dosed orally
Pharmacokinetics (PK) of ZL-82：Vz/F | 24hours
  Estimation of apparent volume of distribution when dosed orally
Pharmacokinetics (PK) of ZL-82：Kel | 24hours
  Estimation of the elimination rate constant of a drug in the body

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lijuan, doctor, Study Chair — West China Hospital
Locations (1):
- Affiliated Hospital of Guizhou Medical University, Guizhou, GuiYang, China

IPD SHARING:
Plan to Share IPD: No